CLINICAL TRIAL: NCT06181630
Title: A Phase IV Postmarketing Study Evaluating Ozanimod Concentrations in the Breast Milk of Lactating Women Receiving Ozanimod Therapeutically
Brief Title: A Lactation Study in Women Receiving Treatment With Ozanimod
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Replaced with another clinical trial
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM047-030
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lactating Women; Breastfed Infants
Keywords: Ozanimod; BMS-986374
MeSH Terms: interventions — Milk, Human; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lactating women receiving treatment with Ozanimod and their infants (Experimental)
  Interventions: Diagnostic Test: Breast milk, plasma, and blood samples

INTERVENTIONS:
Diagnostic Test: Breast milk, plasma, and blood samples — Although this study is non- interventional regarding treatment with ozanimod, the study is considered interventional due to the collection of breast milk and plasma from the lactating women and blood samples from their breastfed infants and the additional diagnostic and monitoring procedures required for the study.

SUMMARY:
The purpose of this study is to assess the concentrations of ozanimod and its major metabolites in breast milk and the effects on breastfed infants.

ELIGIBILITY:
Inclusion Criteria:

* Adult female participant is already planning or currently being treated with ozanimod per the current locally approved prescribing information.
* Adult female participant has delivered a single normal-term infant (at least 37 weeks gestation).
* Adult female participant is at least 2 weeks postpartum but not more than 12 months postpartum by Study Visit 1.
* Infant participant has normal weight for gestational age (above tenth percentile) at birth.

Exclusion Criteria:

* Adult participant is pregnant, planning to become pregnant, or are of childbearing potential and not using an effective contraceptive method.
* Adult participant is not breastfeeding or pumping milk.
* Adult participant has received any live vaccinations within 4 weeks prior to the start of ozanimod treatment.
* Infant participant was born less than 37 weeks gestation

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Average concentration at steady state (Css-avg) in breast milk | Predose; Up to 24 hours post dose
Area under the concentration-time curve over the dosing interval (AUCtau) in breast milk | Predose; Up to 24 hours post dose
Drug daily infant dose | Predose; Up to 24 hours post dose
Drug relative infant dose | Predose; Up to 24 hours post dose

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 5 months
Number of participants with clinical laboratory abnormalities | Up to approximately 5 months
Number of participants with vital sign abnormalities | Up to approximately 5 months
Number of participants with physical examination abnormalities | Up to approximately 5 months
Plasma trough observed plasma concentration at the end of a dosing interval at steady state (Ctrough) | Predose; Up to 12 hours post dose
Maximum observed concentration in breast milk over the dosing interval (Cmax) | Predose; Up to 24 hours post dose
Minimum observed concentration in breast milk over the dosing interval (Cmin) | Predose; Up to 24 hours post dose
Time to reach Cmax (Tmax) | Predose; Up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Las Vegas Clinical Research Unit, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06181630.html